CLINICAL TRIAL: NCT00465868
Title: Magnetic Resonance Imaging, Myocardial Infarction and Development of Heart Failure.
Brief Title: MR, Myocardial Infarct and Heart Failure
Acronym: KoMPiS
Status: Completed | Type: Observational
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Helse Vest (Other); Norwegian Foundation for Health and Rehabilitation (Other); Norwegian Heart and Lung Patient Organization (Unknown); Sparebank 1 SR-Bank Gavefond (Unknown); Amersham Health (Industry)
Responsible Party: Sponsor
Other Study IDs: StaHF461301
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2008-06

CONDITIONS: Heart Failure, Congestive
Keywords: Acute Myocardial Infarction; Coronary Revascularization; Microvascular Obstruction; Cardiac MR; Collagen Turnover; Heart failure, post-mi
MeSH Terms: conditions — Heart Failure | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — collagen markers, inflammatory markers and heart failure markers
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: PCI (percutaneous coronary intervention) — Outcome of PCI following AMI

SUMMARY:
KoMPiS is a contrast aided cardiac magnetic resonance study of microvascular obstruction and left ventricular remodelling following acute revascularised anterior myocardial infarction. The study will monitor the included patients for 12 months following the acute myocardial infarct and collect data from MR scans and blood samples. The study is designed to demonstrate that obstruction of blood flow in the peripheral (small) vessels of the cardiac muscle is an important factor in the post-MI development of left ventricle dysfunction that occurs in many patients, despite of a successful re-opening of the occluded coronary artery that caused the MI.

DETAILED DESCRIPTION:
Introduction. Cardiovascular disease is responsible for 30 % of worldwide mortality, accounting for approximately 15 million deaths per year. Improvement in medical treatment strategies during the last decades has produced a tremendous decrease in mortality in connection with acute myocardial infarction (AMI). Since the 1960's, short-term mortality (30 days) has decreased from approximately 30 % to the current mortality rate of 6,5%. The success of modern treatment of AMI has, however, led to an increasing number of patients surviving AMI, thus creating a growing group of high-risk patients that need further treatment and care. The development of heart failure and the risk of recurrent ischemia and reinfarction are the two main threats to this population. To further improve the treatment and outcomes in this high risk population, early risk stratification based on a thorough understanding of the operating mechanisms behind the transition from acute infarction to heart failure is necessary.

AMI, reperfusion and microvascular obstruction. Reperfusion therapy has been one of the major successes in the treatment of AMI, and there are numerous studies to support the idea of opening occluded coronary arteries, especially in the context of an AMI. However, even in the presence of a patent infarct related artery, there may still be inadequate reperfusion at the tissue level. This phenomenon, known as no-reflow, may preclude optimal reperfusion because of microvascular obstruction. It is estimated that microvascular obstruction occurs in 30-40% of all revascularised patients in spite of a patent artery; the exact underlying pathophysiological mechanisms are partially unknown. Microvascular obstruction may possibly be due to sequestration of neutrophils in the microvasculature that subsequently lead to microvascular occlusion by erythrocytes, leucocytes and cellular debris. It remains unclear whether the stimulus for the development of microvascular obstruction originates during coronary occlusion exclusively or if reperfusion plays an active role in progression of the phenomenon.

Microvascular obstruction and heart failure. The presence of microvascular obstruction following AMI, predicts unfavourable postinfarction prognosis and development of left ventricular dysfunction and left ventricular remodelling. Left ventricular remodelling is associated with development of heart failure and is directly related to the magnitude of microvascular obstruction early after experimental and clinical AMI1, as well as 6 months after the acute event. The mechanisms by which microvascular obstruction induces ventricular remodelling remain unknown. Possibilities include the potentiation of wall thinning and infarct expansion early after infarction, as well as potential impairment of infarct healing, given the association between presence of microvascular obstruction and greater transmural scar formation 6 months after AMI.

Assessment of microvascular obstruction. Until recently, microvascular obstruction could only be assessed by methods such as radioactive micro-spheres and other histopathological techniques, that only could be performed at the terminal phase of an experimental study, and not clinically. However, recent advances in the field of non-invasive cardiac imaging have enabled the serial assessment of this phenomenon by cardiac magnetic resonance imaging (CMR), thereby facilitating a much greater understanding of its pathophysiological and prognostic significance.

Assessment of left ventricular remodelling by CMR. The pathologic changes associated with the development of heart failure include changes in geometry and function, myocytes and extracellular matrix. Assessment of left ventricular remodelling includes estimation of left ventricular size and shape, left ventricular mass and a functional assessment including an estimation of ejection fraction.

Biochemical markers of scar formation, inflammation and LV dysfunction. Prognosis after MI is related both to the extent of myocardial cell-loss and the quality and quantity of repair of the infarcted myocardium. The fate of fibrous tissue following acute myocardial infarction, including regression, persistence or progression of fibrosis is important for the understanding of the underlying mechanisms behind the progressive nature of LV remodelling following AMI. Non-invasive assessment of fibrous tissue formation may be accomplished by measuring serum markers of collagen turnover.

Following AMI, fibrillar collagen appear both in the infarct scar and remote to the site of the myocardial infarction, including viable tissue of the infarcted and noninfarcted ventricles. In rats, procollagen mRNA for collagens type I and III is increased in the right ventricle from day 2 onwards after a transmural left ventricular MI. The increased collagen turnover may last for several months or even years.

Aminoterminal propeptide of type I procollagen (PINP) and aminoterminal propeptide of type III procollagen (PIIINP) are liberated during collagen biosynthesis, and they may be used as markers of this process. PIIINP reflects the turnover of soft tissue collagen and is elevated after AMI, reaching a plateau after four days with the largest increase in patients with large infarctions and acutely reduced LV function. Increased serum PIIINP measured in the subacute phase of myocardial infarction is associated with persistently depressed LV ejection fraction, dilatation and restrictive diastolic filling. Patency of the infarct related artery reduces the PIIINP response and scar formation.

The role of type I collagen following AMI is less clear. It has been suggested that there is a late rise in the synthesis of type I collagen after myocardial infarction, but this remains to be shown. Among patients with heart failure of mixed aetiology (ischemic and non-ischemic), increased levels of CIPT, PINP and PIIINP are associated with an increased risk of death.

The modulation of collagen deposition and scar formation is accomplished by an intricate interplay between neurohormones (eg. aldosterone, angiotensin I and II, bradykinins, catecholamines and natriuretic peptides) and the inflammatory system. The relationship between CMR, collagen markers and neurohormones is not known in this setting.

Study aims. To characterize disease progression and to elucidate the operative pathophysiological mechanisms in patients with evidence of microvascular obstruction on contrast enhanced CMR following acute AMI.

Study plan. This is a single centre observational study, designed to assess differences between patients with and without CMR evidence of microvascular obstruction. To assure a homogenous group of patients, only successfully revascularised patients with AMI caused by a single proximal/mid LAD, CX or RCA occlusion as assessed by coronary angiography, will be included. Only patients with functionally single vessel disease and without former heart disease will be included. Patients will be selected for screening and requested to participate following the acute PCI. The first CMR will be performed at 48±12 hours following the primary PCI. A follow-up CMR will be performed one week, two months and one year following the index PCI. At every CMR examination (including the screening phase), blood samples will be collected, and clinical examination and an echocardiography will be performed. The study population will be managed during and after their AMI according to current optimal guidelines, and all patients will be considered for the same medical therapy, including ACE inhibitors and beta-blockers. The study will evaluate the presence of microvascular obstruction at baseline vs. changes over time in CMR data and biochemical markers of collagen turnover, neurohormonal activity and inflammation.

Sample size estimation. To detect a difference in LV mass of 10g with a power of 80% and a p = 0,05, it is necessary to include 14 patients. To show a difference in ejection fraction of 5% with a power of 90% and p = 0,05, it is sufficient to include 5 patients. In a study by Wu and coworkers, late enhancement CMR demonstrated a significant difference in clinical outcome following myocardial infarction when 38 patients (with or without congestive heart failure) were divided into three groups according to the size of infarction. To account for dropout and biological variation we will include a minimum of 20 patients with microvascular obstruction. It is estimated that microvascular obstruction persists in around 30-40% of all patients undergoing revascularisation. The group of patients without microvascular obstruction will consequently be 40 patients, generating a total study population of 60 patients.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > 18 years of age, non-child bearing potential
* First time acute myocardial infarction, as determined by evidence of transmural ischemia in the ECG and a rise in cardiac-Troponin-T (TNT) > 0,1 (μg/l), followed by
* A successful acute PCI of a single vessel disease with a proximal/mid left anterior descent artery (LAD), circumflex artery (RCX) or right coronary artery (RCA) lesion (the index PCI).

Exclusion Criteria:

* Extensive cardiopulmonary resuscitation.
* Haemodynamically unstable patients, unable to leave the coronary care unit for the CMR examination.
* Use of fibrinolytics immediately prior to the index PCI.
* Significant primary valve disease,
* Autoimmune disease causing an increase in collagen turnover
* Active cancer disease
* Need for immunosuppressive treatment,
* Significantly reduced liver function
* Contraindications for performing a cardiac MRI-scan (claustrophobia, and implanted ferromagnetic devices, known allergic reactions to Omniscan™).
* Inability to understand the consent form or cooperate during the 1 year follow up.
* Comorbidity with poor prognosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admited with AMi and rescue PCI.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2004-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Dickstein, PhD, Study Chair — Universiy of Bergen, Norway
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

REFERENCES:
- [Derived] Manhenke C, Ueland T, Jugdutt BI, Godang K, Aukrust P, Dickstein K, Orn S. The relationship between markers of extracellular cardiac matrix turnover: infarct healing and left ventricular remodelling following primary PCI in patients with first-time STEMI. Eur Heart J. 2014 Feb;35(6):395-402. doi: 10.1093/eurheartj/eht482. Epub 2013 Nov 18. PMID 24255130
- [Derived] Orn S, Manhenke C, Greve OJ, Larsen AI, Bonarjee VV, Edvardsen T, Dickstein K. Microvascular obstruction is a major determinant of infarct healing and subsequent left ventricular remodelling following primary percutaneous coronary intervention. Eur Heart J. 2009 Aug;30(16):1978-85. doi: 10.1093/eurheartj/ehp219. Epub 2009 Jun 6. PMID 19502624
- [Derived] Orn S, Manhenke C, Ueland T, Damas JK, Mollnes TE, Edvardsen T, Aukrust P, Dickstein K. C-reactive protein, infarct size, microvascular obstruction, and left-ventricular remodelling following acute myocardial infarction. Eur Heart J. 2009 May;30(10):1180-6. doi: 10.1093/eurheartj/ehp070. Epub 2009 Mar 19. PMID 19299430